CLINICAL TRIAL: NCT03415854
Title: A Phase II Pilot Trial Of Paclitaxel Protein Bound Plus Cisplatin Plus Gemcitabine and the Addition Of Paricalcitol Upon Disease Progression in Patients With Previously Untreated Metastatic Pancreatic Ductal Adenocarcinoma (NABPLAGEMD)
Brief Title: Paclitaxel Protein Bound Plus Cisplatin Plus Gemcitabine and Paricalcitol for Pancreatic Adenocarcinoma (NABPLAGEMD)
Acronym: NABPLAGEMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Collaborators: Barts Cancer Institute (Other); Abramson Cancer Center at Penn Medicine (Other); Salk Institute for Biological Studies (Other); Mayo Clinic (Other); Princeton University (Other); Imaging Endpoints (Unknown); Translational Genomics Research Institute (Other); Stand Up To Cancer (Other); Cancer Research UK (Other); Lustgarten Foundation (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU2C HRI NPG-001
Record Dates: First submitted 2018-01-09; First posted 2018-01-30 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma; Pancreatic Adenocarcinoma; Pancreas Metastases; Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — paricalcitol; Cisplatin; Taxes; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Paricalcitol (Zemplar) (Experimental): Participants will be treated with the regimen according to the study protocol. Participants will complete 3 cycles (cycle is 21 days) and then will be evaluated for CA19-9 normalization and undergo imaging to determine response, if any.
  Interventions: Drug: Paricalcitol (Zemplar)

INTERVENTIONS:
Drug: Paricalcitol (Zemplar) — combination therapy
  Other Names: Cisplatin (Platinol); Paclitaxel Protein Bound (Abraxane); Gemcitabine (Gemzar)

SUMMARY:
The purpose of this study is to determine if the combination of paclitaxel protein bound, gemcitabine, cisplatin, paricalcitol are effective in individuals with previously untreated metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer continues to be a highly lethal disease with an overall 5 year survival of only 8%. Since 2004, the incidence of pancreatic cancer has been increasing by 1.5% per year and it is estimated that there will be 53,670 new cases diagnosed in the United States in 2017, with 43,090 expected deaths. Pancreatic cancer is the third most common cause of cancer-related deaths in both men and women, and the incidence is about equal in both sexes. Of all types of pancreatic cancers, pancreatic ductal adenocarcinoma (PDA) is by far the most common, representing 80% of cases. Due to lack of adequate screening techniques, greater than 80% of patients at the time of diagnosis present with unresectable, advanced disease. Standard treatment options for inoperable patients with locally advanced and metastatic PDA have been quite limited. Gemcitabine monotherapy, approved by the Food and Drug Administration (FDA) in 1996, demonstrated a median survival of 5.7 months, and has been the mainstay in treating patients with PDA. The first combination regimen to demonstrate any survival benefit compared with gemcitabine alone was gemcitabine plus erlotinib, with median survival of 6.24 months versus 5.91 months for single agent gemcitabine.

A meta-analysis of randomized trials by Heinemann and colleagues showed that patients with advanced pancreatic cancer and a good performance status may benefit from combination chemotherapy with gemcitabine plus a platinum agent or a fluoropyrimidine. Multiple combination regimens are being utilized.

Recently, the regimen of 5-fluorouracil/leucovorin/irinotecan/oxaliplatin (FOLFIRINOX) compared with gemcitabine demonstrated improvement in both progression-free survival (PFS, 6.4 vs. 3.3 months) and overall survival (OS, 11.1 vs. 6.8 months) for patients with a good performance status. FOLFIRINOX, however, is associated with substantial grade 3 and 4 toxicities, including diarrhea, nausea, vomiting, fatigue, neutropenia and febrile neutropenia, and cannot be given to patients >76 years of age or in some cases patients with head of the pancreas tumors. An international phase III trial comparing paclitaxel protein bound (now called paclitaxel protein bound) plus gemcitabine to gemcitabine single agent demonstrated a statistically significant improvement in OS (8.5 vs. 6.7 months) for advanced pancreatic cancer patients using the gemcitabine and paclitaxel protein bound over gemcitabine alone.

A recently completed phase Ib/II trial of the combination of paclitaxel protein bound plus gemcitabine plus cisplatin in previously untreated stage IV pancreatic adenocarcinoma patients was presented at the 2017 Gastrointestinal Cancer Symposium. In 24 patients with stage IV pancreatic cancer they reported 8.3% complete response (CR), 62.5% partial response (PR), 16.7% stable disease and 12.5% progressive disease. The rationale for adding cisplatin to paclitaxel protein bound and gemcitabine is that in a study of 1,029 patients whose pancreatic cancer tumors underwent molecular profiling, 57% of these tumors were negative for expression of the excision repair cross-complementation group 1 (ERCC1), indicating sensitivity to a platinum anti-tumor agent. In addition to the above, in our whole genome/transcriptome sequencing analysis, we found that abnormal repair pathways were a feature of all of the pancreatic cancers that were sequenced. Cisplatin prevents cellular deoxyribonucleic acid (DNA) repair by binding to and causing crosslinking of DNA, triggering apoptosis. Cisplatin has been used in other combination regimens to treat patients with PDA. For example, the cisplatin, epirubicin, 5-fluorouracil and gemcitabine (PEFG) regimen had an acceptable toxicity profile and was associated with a 24% partial response rate, 5 month PFS and 8.3 month OS as second line therapy.

Most recently, a study showed that Vitamin D can change the pancreatic tumor microenvironment from an immunologically suppressive (tumor promoting) one to an immunologically hostile one (e.g. decreased IL-6, decreased CXCL12 etc.). In addition, in the same study, the vitamin D ligand calcipotriol decreased production of collagen, decreased myeloid derived suppressor cells (MDSCs) and decreased regulatory T cells. Remarkably, in clinical practice, the vitamin D analogue paricalcitol was observed to reverse chemotherapy resistance. Two individuals with pancreatic adenocarcinoma who were receiving paclitaxel protein bound and gemcitabine based combination chemotherapy developed progressive disease which was reversed by the addition of paricalcitol.

Based upon these promising clinical and pre-clinical data we are initiating a clinical trial combining paclitaxel protein bound, gemcitabine, and cisplatin for patients with metastatic PDA. When these patients develop progressive disease the vitamin D analog paricalcitol will be added to the regimen. The treatment will continue until further disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age; male or female.
2. Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma.
3. Capable of providing informed consent and complying with trial procedures including obtaining paired biopsies during therapy
4. Karnofsky Performance Status (KPS) of ≥ 70%.
5. Life expectancy ≥ 12 weeks.
6. Measurable tumor lesions according to RECIST 1.1 criteria.
7. Women must agree not to become pregnant (e.g. post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study and until 90 days after last dose of study treatment. Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating. Both male and female patients of reproductive potential must agree to use a reliable method of birth control during the study.

Exclusion Criteria:

1. Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatments in the adjuvant setting with gemcitabine and/or Fluorouracil (5-FU) or gemcitabine administered as a radiation sensitizer are allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
2. Palliative surgery and/or radiation treatment less than 4 weeks prior to initiation of study treatment.
3. Exposure to any investigational agent within 4 weeks prior to initiation of study treatment.
4. Evidence of central nervous system (CNS) metastasis (negative imaging study, if clinically indicated, within 4 weeks of Screening Visit).
5. History of other malignancies (except cured basal or squamous cell carcinoma, superficial bladder cancer, prostate cancer in active surveillance, or carcinoma in situ of the cervix) unless documented free of cancer for ≥2 years.
6. Laboratory values: Screening serum creatinine >1.5 mg/dL; total bilirubin > (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 2.5x ULN or ≥ 5.0×ULN if liver metastases are present; absolute neutrophil count <1,500/mm3, platelet concentration <100,000/mm3, hematocrit level <27% for females or <30% for males, or coagulation tests (prothrombin time [PT], partial thromboplastin time [PTT], International Normalized Ratio [INR]) >1.5×ULN unless on anticoagulation agents.
7. Current, serious, clinically significant cardiac arrhythmias as determined by the investigator.
8. History of HIV infection.
9. Active, clinically significant serious infection requiring treatment with antibiotics, antivirals or anti-fungals.
10. Any condition that might interfere with the patient's participation in the study or in the evaluation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate | At the end of 3 cycles (each cycle is 21 days)
  Participants will have an MRI completed after 3 cycles to determine if the tumor has responded to treatment. RECIST 1.1 criteria will be used to evaluate response. A confirmatory positron emission tomography (PET) scan may be ordered to confirm complete response.

SECONDARY OUTCOMES:
Carbohydrate Antigen 19-9 (CA19-9) value | At the end of each cycle (each cycle is 21 days)
  Laboratory testing will be used to determine if the CA19-9 value has normalized after each cycle of treatment.
changes in circulating biomarkers induced by paricalcitol | At the end of each cycle (each cycle is 21 days)
  Laboratory testing will be used to determine any changes in circulating biomarkers induced by paricalcitol. Biomarkers to be tested include: Stromal content (collagen and hyaluronan), CD31 (cluster of differentiation 31) staining, PD-1(programmed cell death-1) / PDl-1 (protein disulfide isomerase) staining and expression, IHC (Immunohistochemistry) evaluation of key immune cell populations (cytotoxic T Cells, TAMs (tumor-associated macrophages), MDSCs (myeloid-derived suppressor cells), and Tregs (regulatory T cells in cancer)), clonality of intra-tumoral T cells by TSR (tumor stroma ratio) sequencing (a measure of intratumoral response), expression of VDR (vitamin D receptor) regulated inflammatory gene (IL6 (interleukin 6), CXCL1 (chemokine (C-X-C motif) ligand 1), CSF2 (colony stimulating factor 2), CXCLR(chemokine (C-X-C motif) receptor)), VDR and CYP24A1 (cytochrome P450 family 24 subfamily A member 1), mutational and transcriptional profile.
changes in circulating biomarkers induced by chemotherapy | At the end of each cycle (each cycle is 21 days)
  Laboratory testing will be used to determine any changes in circulating biomarkers induced by chemotherapy. Biomarkers to be tested include: Stromal content (collagen and hyaluronan), CD31 (cluster of differentiation 31) staining, PD-1(programmed cell death-1) / PDl-1 (protein disulfide isomerase) staining and expression, IHC (Immunohistochemistry) evaluation of key immune cell populations (cytotoxic T Cells, TAMs (tumor-associated macrophages), MDSCs (myeloid-derived suppressor cells), and Tregs (regulatory T cells in cancer)), clonality of intra-tumoral T cells by TSR (tumor stroma ratio) sequencing (a measure of intratumoral response), expression of VDR (vitamin D receptor) regulated inflammatory gene (IL6 (interleukin 6), CXCL1 (chemokine (C-X-C motif) ligand 1), CSF2 (colony stimulating factor 2), CXCLR(chemokine (C-X-C motif) receptor)), VDR and CYP24A1 (cytochrome P450 family 24 subfamily A member 1), mutational and transcriptional profile.
pharmacodynamics effect of Paricalcitol | At the end of 2 cycles (each cycle is 21 days)
  Tumor biopsy testing will be used to determine the pharmacodynamics effect of Paricalcitol for patients with metastatic PDA (pancreatic ductal adenocarcinoma) . Fresh tumor biopsies will be obtained to evaluate the pharmacodynamics effect of Paricalcitol on PDA, a core biopsy will be performed at baseline prior to the addition of paricalcitol along with one after 2 cycles of the triplet regimen plus paricalcitol (6 weeks).
Parathyroid Hormone (PTH) | At the end of each cycle (each cycle is 21 days)
  Laboratory testing will be used to monitor any changes in parathyroid hormone (PTH) in individuals treated with paricalcitol.
Vitamin D 25-hydroxy (OH) | At the end of each cycle (each cycle is 21 days)
  Laboratory testing will be used to monitor and measure the serum levels of Vitamin D 25-OH after each cycle of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Erkut Borazanci, MD, Principal Investigator — HonorHealth Research Institute
Locations (1):
- HonorHealth Research Institute, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
If the study site is a 'covered site' under the definitions of the Health Insurance Portability and Accounting Act (HIPAA), the Investigator will ensure that the patient consents to the use of data by HonorHealth and its designees for the purposes of regulatory submissions, study publications, and drug approval.
  Stand Up To Cancer (SU2C) will be notified of any outputs of the research such as guidelines, publications, presentation, changes in service delivery etc. prior to external submission or presentation. In any oral or written report or poster presentation of Results or otherwise relating to the Research, the support of Cancer Research UK (CRUK), SU2C and the Lustgarten foundation will be acknowledged, displaying the relevant logs where possible. Any publications resulting from research funded in whole or in part by the Grant must be cited as required per signed confidentiality agreements.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: To be determined
Access Criteria: The Investigator and any other study personnel involved in this study shall not disclose, or use for any purposes (other than for the performance of this study), any data, records, or other information (hereinafter collectively "information") disclosed to the Investigator or other study personnel. Such information shall remain the confidential and proprietary property of HonorHealth, and shall be disclosed only to the Investigator or other designated study personnel.
  The obligation of non-disclosure shall not apply to the following:
  * relevant disclosure to potential study participants for the purpose of obtaining informed consent;
  * information after such time that it is or becomes publicly available through no fault of the Investigator or other study personnel; and,
  * information after such time that it is disclosed to the Investigator by a third party entitled to disclose such information.